CLINICAL TRIAL: NCT02799394
Title: Effect of Activity Modification and Exercises in Young Adolescents With Osgood Schlatter Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Michael Skovdal Rathleff, Senior Researcher, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N- 20140100-1
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Osgood Schlatter Disease
MeSH Terms: conditions — Osteochondrosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Activity modification, exercises and gradual return to sport (Experimental)
  Interventions: Other: Activity modification, exercises and gradual return to sport

INTERVENTIONS:
Other: Activity modification, exercises and gradual return to sport

SUMMARY:
The purpose of this study is to investigate the effect of activity modification, exercises and a gradual return to sport in adolescents (age 10-14) with Osgood Schlatter disease. The primary outcome is self-reported recovery on a 7-point Likert scale at 3 months. Secondary endpoints include 4 and 8 weeks and 6 and 12 months after inclusion into the project. The adolescents will be recruited from primary schools, general practitioners and through online advertising on Facebook.

ELIGIBILITY:
Inclusion Criteria:

* 10-14 years of age
* Pain at tuberositas patellae during two or more of the following activities: Sitting with a bent knee, squatting, running, jumping or stair ambulation
* Pain during palpation of tuberositas patellae
* Knee pain for 6 weeks or more

Exclusion Criteria:

* Other knee conditions that may manifest as anterior knee pain (Patellofemoral pain, iliotibial band syndrome, sinding-larson-johanson disease).
* Previous surgery
* Pain from the hip or back that interferes with activities of daily living.
* Habitual patella luxations
* Clinical suspicion of meniscal lesion

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Self-reported recovery on a 7-point Likert scale | 3 months

SECONDARY OUTCOMES:
Self-reported recovery on a 7-point Likert scale | 4 and 8 weeks + 6 and 12 months after inclusion.
Self-report questionnaire "Knee Injury and Osteoarthritis Outcome Score" | 4, 8 and 12 weeks + 6 and 12 months after inclusion.
Isometric hip and knee extension strength assessed using a strap-mounted dynamometer | 4, 8 and 12 weeks after inclusion.
Pressure pain thresholds at tuberositas patella, center of patella and lateral elbow assessed by a hand held pressure algometer. | 4, 8 and 12 weeks after inclusion.
Thigh circumference measured using tape measure. | 4, 8 and 12 weeks after inclusion.
Vertical jump for height [calculated as the difference between reach height and maximal jump height. This will be measured using a ruler] | 4, 8 and 12 weeks after inclusion.
Single leg jump for distance (defined as the maximal length the subject can jump on one leg. Measured using a ruler). | 4, 8 and 12 weeks after inclusion.
Flexibility of the hamstrings and quadriceps [measured using goniometer]. | 4, 8 and 12 weeks after inclusion.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aalborg Universitetshospital, Aalborg, The North Denmark Region
  - Hvidovre-Amager Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes
Data will be made publicly available no later than six months after the final publication.

REFERENCES:
- [Derived] Rathleff MS, Winiarski L, Krommes K, Graven-Nielsen T, Holmich P, Olesen JL, Holden S, Thorborg K. Activity Modification and Knee Strengthening for Osgood-Schlatter Disease: A Prospective Cohort Study. Orthop J Sports Med. 2020 Apr 6;8(4):2325967120911106. doi: 10.1177/2325967120911106. eCollection 2020 Apr. PMID 32284945